CLINICAL TRIAL: NCT02495298
Title: Evaluation of Fascial Manipulation for the Conservative Treatment of Carpal Tunnel Syndrome: Double Blind Randomized Clinical Trial, Phase II
Brief Title: Fascial Manipulation on the Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marta Imamura (Other)
Responsible Party: Sponsor-Investigator, Marta Imamura, Coordinator of the Clinical Trial Site of the Institute of Physical Medicine and Rehabilitation Medicine of HCFMUSP, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fascial Manipulation on CTS
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Fascial manipulation; Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Fascial Manipulation (Experimental): Seven patients with diagnosis of CTS, received five sessions of Fascial Manipulation performed by a physiotherapist. The sessions were performed once a week, and each session were 30 to 45 minutes long as to cover different painful spots.
  Interventions: Procedure: Fascial Manipulation
- Placebo Fascial Manipulation (Sham Comparator): Seven patients with diagnosis of CTS, received five sessions of Sham Fascial Manipulation performed by a physiotherapist. The sessions were performed once a week, and each session were 30 to 45 minutes long as to cover different painful spots.
  Interventions: Procedure: Sham Fascial Manipulation

INTERVENTIONS:
Procedure: Fascial Manipulation — The Fascial Manipulation was performed by a physiotherapist on the spots indicated by clinician as the most painful ones due to CTS. The selected spots were informed to the physiotherapist after the clinical anamnesis.
  Arms: Treatment Fascial Manipulation
Procedure: Sham Fascial Manipulation — After the clinical anamnesis, a physiotherapist performed the Fascial Manipulation on different spots, rather than the spots the clinician considered the most painful ones due to CTS.
  Arms: Placebo Fascial Manipulation

SUMMARY:
The trial aims to evaluate the effectiveness of Fascial Manipulation on pain reduction, functional recovery and nerve conduction of patients with Carpal Tunnel Syndrome (CTS). Visual Analogue Scale (VAS), Disabilities of the Arm, Shoulder and Hand scale (DASH), Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and Electroneuromyography were assessed.

The study is blind for the patient and the raters.

DETAILED DESCRIPTION:
This is a prospective, randomized, placebo controlled, rater blind trial to evaluate the effectiveness of Fascial Manipulation as a therapy for CTS. Fascial Manipulation is an intense friction performed by the elbows or the distal extremities of the interphalangeal articulation of the index finger for some minutes as to promote hyperemia to restore the collagen fibers ability to slide against each other. The friction lasts from 2 to 4 minutes.

In this trial, 14 patients were randomized in two groups: The intervention group received fascial manipulation for CTS and the other group, received fascial manipulation on spots not related to CTS. This last group was the placebo control group.

The treatment was performed once a week for 5 weeks consecutively and the follow up visits for the assessments were performed 10 days and 3 months after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* CTS degrees Ia, Ib and II diagnosis according to clinical evaluation and electroneuromyography;
* Wrist and finger paresthesia for more than 3 months prior to screening visit;
* Moderate to intense pain: VAS>4.
* Ability to understand and respond to the questionnaires used in the trial;
* Ability to understand the Informed Consent Form;
* Sign the Informed Consent Form.

Exclusion Criteria:

* Psychiatric disorders;
* Fibromyalgia;
* Rheumatologic diseases;
* Other conditions related to CTS, as renal failure, diabetes, acromegaly, hyperthyroidism, multiple myeloma;
* History of neoplasia;
* History of surgery at Carpal Tunnel;
* History of use of illegal drugs;
* History of chronic use of corticosteroids;
* Corticosteroid infiltration one month prior to inclusion in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the VAS score for pain at 10 days after the end of the treatment. | Baseline and 10 days after end of the treatment.

SECONDARY OUTCOMES:
Change from baseline in pain on the VAS score for pain at 3 months after the end of the treatment. | Baseline and 3 months after end of the treatment.
Change from baseline in function on BCTQ score for function at 10 days and 3 months after the end of the treatment. | Baseline, 10 days and 3 months after the treatment
  The Boston Carpal Tunnel Syndrome Questionnaire is a self rated evaluation which assesses the function, with 8 items, and the symptoms, with 11 items, of patients with CTS. Each item is a 5-point scale.
Change from baseline in function on DASH score for function at 10 days and 3 | Baseline, 10 days and 3 months after the treatment
  The DASH scale is a self rated evaluation for upper limbs which assesses symptoms and function with 30 items in total. Each arm has a score from 1 to 5, in which highest score indicates highest incapacities.
Change from baseline in nerve conduction on Electroneuromyography test for nerve conduction at 10 days after the end of the treatment | Baseline and 10 days after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, MD, Principal Investigator — Instituto de Medicina Física e Reabilitação HCFMUSP
Locations (1):
- Instituto de Medicina Fisica e Reabilitacao HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No